CLINICAL TRIAL: NCT03423719
Title: Effect of a 16-week Supplementation With a Mediterranean Fruit and Vegetables Extract Rich in Polyphenols, Fiit-ns®, on Health-related Quality of Life of Overweight and Obese Volunteers: a Randomized, Double-blind, Parallel Trial
Brief Title: Evaluation of Fiit-ns® in Health-related Quality of Life Improvement in Overweight and Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fytexia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FITCT2015
Record Dates: First submitted 2018-01-30; First posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): This arm receives 2 x 450 mg capsules of Fiit-ns®, a blend of polyphenol-rich fruit and vegetables extracts, daily for 16 weeks.
  Interventions: Dietary Supplement: Fiit-ns®
- Placebo (Placebo Comparator): This arm receives 2 x 450 mg capsules of Placebo, containing maltodextrin only, daily for 16 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fiit-ns® — Fiit-ns® is a blend of polyphenol-rich extracts from grapefruit, grape, green tea, guarana and black carrot. It also provides Vitamin B3. Daily dosage is 900 mg in two 450 mg-capsules for 16 weeks.
  Arms: Verum
Dietary Supplement: Placebo — Placebo product is 100% maltodextrin. Daily dosage is 900 mg in two 450 mg-capsules of identical appearance than the supplement capsule for 16 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of a 16-week supplementation with a polyphenol-rich extract, Fiit-ns®, on improvement of health-related quality of life (HR-QOL) of overweight and obese volunteers, as compared to placebo. Previous beneficial results from a pilot study showed that the supplementation may improve quality of life as well as body composition. Based on such results, this pivotal study is statistically powered to detect significant differences in HR-QOL assessed with the Short Form-36 Health survey (SF-36) between baseline (Week 1, W1) and end of the supplementation period (Week 16, W16).

ELIGIBILITY:
Inclusion Criteria:

* 25 kg/m2 ≤ Body Mass Index (BMI) ≤ 40 kg/m2
* 25-55 years old

Exclusion Criteria:

* Metabolic and/or chronic disease (diabetes, dyslipidemia, thyroiditis, inflammatory disease, immunological disease, asthma, anxiety, depression)
* Allergy to one of the ingredients of the supplement
* Current involvement of involvement within the 6 previous months in a chronic supplement program, chronic treatment program, weight loss program
* Smoking cessation
* High alcohol consumption
* Pregnancy
* Breastfeeding
* Menopausal women
* Involvement in physical activity more than twice a week

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in health-related quality of life as assessed by the SF-36 Health Survey | Baseline (Week 1) and end of the supplementation period (Week 16)

SECONDARY OUTCOMES:
Change in body weight | Baseline (Week 1) and end of the supplementation period (Week 16)
  Change in body weight is measured with calibrated weighing scales
Change in waist circumference | Baseline (Week 1) and end of the supplementation period (Week 16)
  Change is waist circumference is measured with a non-stretchable tape and used to calculate change in Index of Central Obesity (ICO)
Change in total body fat mass | Baseline (Week 1) and end of the supplementation period (Week 16)
  Change in total body fat mass is measured with Dual-Energy X-ray Absorptiometry (DXA) scan
Change in trunk fat mass | Baseline (Week 1) and end of the supplementation period (Week 16 )
  Change in trunk fat mass is measured with Dual-Energy X-ray Absorptiometry (DXA) scan
Change in physical activity level | Baseline (Week 1) and end of the supplementation period (Week 16)
  Physical activity is assessed with International Physical Activity Questionnaire (IPAQ) IPAQ consists in 27 items that cover 4 different domains of physical activity (working, transportation, housework and gardening & leisure-time) in terms of time spent during the 7 previous days.
  Total score is the sum of the 4 domains and results are presented as an estimation of energy expenditure in metabolic equivalent-minutes per week (Met-min/week).

CONTACTS AND LOCATIONS:
Overall Officials: Pedro E Alcaraz Ramon, Principal Investigator — UCAM (Universidad Catolica San Antonio de Murcia)
Locations (1):
- UCAM (Universidad Catolica San Antonio de Murcia), Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided